CLINICAL TRIAL: NCT05647395
Title: Effects of Different Deflation Methods on Coughing Response and Hemodynamics During Extubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20221121
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Deflating Method
Keywords: Deflating method; Extubation phase; Coughing reaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slowly and evenly draw the gas in the cuff (Experimental)
  Interventions: Behavioral: Tracheal tube cuffs differ in deflation
- One-time aspiration of tracheal catheter cuff gas (No Intervention)

INTERVENTIONS:
Behavioral: Tracheal tube cuffs differ in deflation — When removing the endotracheal tube, the gas in the cuff is drawn at a uniform and slow pace
  Arms: Slowly and evenly draw the gas in the cuff

SUMMARY:
Patients with endotracheal intubation and general anesthesia often have severe choking and hemodynamic fluctuations during the extubation period, which increases the risk of cerebrovascular accident, arrhythmia, incision bleeding and so on . This study aimed to observe the effects of different methods of deflating of endotracheal tube cuffs on cough response and hemodynamics during periextubation in patients undergoing general anesthesia surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Elective endotracheal intubation under general anesthesia.
2. Operation time < 3 h.
3. ASA grade I or II.
4. Age 18~65 years old.

Exclusion Criteria:

1. Throat and neck surgery.
2. Those assessed to have a high risk of reflux aspiration.
3. Difficulty intubation.
4. History of snoring before surgery.
5. Recent respiratory illness such as chronic cough.
6. Previous airway hyperresponsiveness, such as asthma.
7. recent use of cough suppressants.
8. Patients with severe heart, liver and kidney diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Grading of cough reaction | During extubation procedure
  Grading of cough reactions
Change in Blood pressure | Preoperatively, immediately before extubation, immediately after extubation, 1 minute after extubation, 3 minutes after extubation, 10 minutes after extubation
  Hemodynamics
Change in Heart rate | Preoperatively, immediately before extubation, immediately after extubation, 1 minute after extubation, 3 minutes after extubation, 10 minutes after extubation
  Hemodynamics

SECONDARY OUTCOMES:
Adverse reactions | Within 24 hours after removal of the endotracheal tube
  Hypoventilation, pharyngeal discomfort, hoarseness

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China